CLINICAL TRIAL: NCT04352595
Title: Assess Hemay808 Concentration of Different Dosage Regimen for Mild and Moderate Atopic Dermatitis Patients the Safety and Efficacy of Multicenter, Randomized, Blinded, Excipient Parallel-group Phase Ⅱ Clinical Study
Brief Title: A Phase Ⅱ Study of Hemay808 for Atopic Dermatitis Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Hemay Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Organization: Ganzhou Hemay Pharmaceutical Co., Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HM808AD2S01
Record Dates: First submitted 2020-03-20; First posted 2020-04-20 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 1% Hemay808 (Experimental)
  Interventions: Drug: Hemay808
- 3% Hemay808 (Experimental)
  Interventions: Drug: Hemay808
- 7% Hemay808 (Experimental)
  Interventions: Drug: Hemay808
- vehicle (Placebo Comparator)
  Interventions: Drug: Hemay808

INTERVENTIONS:
Drug: Hemay808 — Hemay808 is a onitment of Hemay028, a small molecule PDE4 inhibitor.

SUMMARY:
Assess Hemay808 concentration of 1%/3%/7% for treatment of mild and moderate adult atopic dermatitis patients.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old and ≤65 years old, gender is not limited;
* It met the diagnostic criteria for atopic dermatitis (AD) of Hanifin&Rajka, and the history of AD before screening was ≥6 months;
* The investigator's overall score (IGA) at the screening period/baseline visit was 2-3;
* The skin lesion area of atopic dermatitis (excluding scalp lesions) is 3%-20% of body surface area (BSA) and suitable for local treatment;
* During the study period and within 3 months after the last administration, fertile female subjects and male subjects who did not receive vasectomy were required to take effective contraceptive measures;
* Those who have full knowledge of the test, participate in the test voluntarily and sign the informed consent.

Exclusion Criteria:

* The lesion area of AD is infected and requires local or systematic treatment with anti-infective drugs, or external administration of strong or potent glucocorticoids (see annex 4) or systematic administration of glucocorticoids to control AD Useing of systemic glucocorticoids and/or immunosuppressants within 4 weeks; Or sunbathing, phototherapy (including ultraviolet therapy, photochemotherapy, etc.); Or systematic use of traditional Chinese medicine or natural medicine for the purpose of treating atopic dermatitis;
* The AD lesion area was marked, tattooed, or hyperpigmented, and was judged by the investigator to interfere with the evaluation of the response to the study's drug therapy;
* Previous use of systemic or local pde-4 inhibitors;
* Suffering from clinically significant active systemic infections;
* 2 times the normal upper limit of ALT or AST >, or the normal upper limit of Cr and > of renal function (study allowed 1 reexamination, excluded if still not meeting the inclusion requirements);
* Unwilling to limit their excessive uv exposure during the study period (e.g., sunbathing and/or tanning devices);
* Received the following treatment in the limited time period prior to baseline evaluation:

  1. . Received biologic therapy (including intravenous immunoglobulin) within 12 weeks or 5 half-lives, whichever is greater;
  2. . Use of systemic glucocorticoids and/or immunosuppressants within 4 weeks; Or sunbathing, phototherapy (including ultraviolet therapy, photochemotherapy, etc.); Or systematic use of traditional Chinese medicine or natural medicine for the purpose of treating atopic dermatitis;
  3. . The following treatment was administered within 2 weeks: systemic anti-infective drugs (both oral and intravenous); Or local use of glucocorticoid or local use of calcineurin inhibitor; Local use of traditional Chinese medicine or natural medicine for the purpose of treating atopic dermatitis; Or other topical drugs for the treatment of atopic dermatitis [zinc oxide oil (paste), black bean oil ointment, doxepin cream, etc.];
  4. . Local anti - microbial preparation was used within 1 week;
* Suffering from serious diseases of the central nervous system, cardiovascular system, respiratory system, liver, kidney, gastrointestinal system, urinary system, endocrine system or blood system, and the researcher believes that may confused result or affect the safety of the subjects;
* Suffering from a serious mental illness or other condition that affects research compliance and may interfere with the conduct of clinical trials;
* A history of malignant tumor;
* With a history of severe allergic reactions to skin topical preparations (including angioedema, allergic reactions, etc.) or known allergic reactions to Hemay808 accessories;
* Screening people who had a long history of drug abuse or alcohol abuse in the first 6 months;
* Female subjects who are suspected to be pregnant, lactating or preparing for pregnancy during the test;
* The subject plans to undergo surgery requiring hospitalization or surgery during his or her participation in the study;
* Those who participated in clinical studies of other drugs/devices and used experimental drugs/devices within the last 3 months of randomized enrollment;
* Other conditions made the researchers considered inappropriate for the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2020-04-24 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-04-02 (Actual)

PRIMARY OUTCOMES:
The change in the EASI score relative to the baseline. | Day 29
  EASI Clinical Signs Severity Sum Score change from Baseline at Day 29

SECONDARY OUTCOMES:
The percentage of subjects achieving Investigator's Global Score (IGA) response which improvement ≥ 2 from baseline. | Day 8, Day 15, Day 22, Day 28
  The IGA is a validated assessment instrument used in clinical studies to rate the severity of AD globally.
The percentage of subjects achieving Investigator's Global Score (IGA) score 0-1. | Day 8, Day 15, Day 22, Day 28
  The IGA is a validated assessment instrument used in clinical studies to rate the severity of AD globally.
The change in the IGA score relative to the baseline. | Day 8, Day 15, Day 22, Day 28
  Change From Baseline in the IGA Clinical Signs Severity Sum Score.
The percentage of subjects achieving EASI90, EASI75, EASI50. | Day 8, Day 15, Day 22, Day 28
  EASI Clinical Signs Severity Sum Score ≥50%, 75%, 90% improvement from baseline.
Absolute change in weekly average of daily peak Pruritus Numerical Rating Scale (NRS). | Day 8, Day 15, Day 22, Day 28
  Range of 0 (No itch) to 10 (Worst imaginable itch)
Change From Baseline in Dermatology Life Quality Index (DLQI) Total Score. | Day 8, Day 15, Day 22, Day 28
  The DLQI is a general dermatology questionnaire that consists of 10 items that assess participant health-related quality of life (daily activities, personal relationships, symptoms and feelings, leisure, work and school, and treatment). It has been extensively used in clinical trials for AD. The DLQI is a psychometrically valid and reliable instrument that has been translated into several languages, and the DLQI total scores have been shown to be responsive to change. The minimally important difference for the DLQI has been estimated as a 2-5 point change from baseline. Each item is scored as "very much (3)", "a lot (2)", "a little (1)" and "not at all (0)". The score can range from 0 to 30. The higher values represent the worse dermatology life quality
The percentage of AD invoved BSA (body surface area) change From Baseline. | Day 8, Day 15, Day 22, Day 28
  AD invoved body surface area.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Dermotology hospital, Chinese academy of medical science, Nanjing, Jiangsu
  - Ningbo second hospital, Ningbo, Zhejiang

IPD SHARING:
Plan to Share IPD: No